CLINICAL TRIAL: NCT00265460
Title: Phase 2 Study of Smoke Free Tobacco and Group Support for Smoking Cessation
Brief Title: Smoking Cessation in Groups and With Tobacco Pastils
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tonga.2005.00.
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Smoking
Keywords: smoking cessation,; nicotine,; smokeless tobacco,; cigarettes
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use | interventions — Tobacco Products

INTERVENTIONS:
Drug: Oliwer Twist smokeless tobacco (tobacco)

SUMMARY:
The purpose of this trial is to examine if smokeless tobacco combined with group support might increase smoking cessation rate compared with groups support in smokers.

DETAILED DESCRIPTION:
The purpose of this trial is to examine if smokeless tobacco (Oliwer Twist) combined with group support (15-20 per group) might increase smoking cessation rate compared with groups support cold turkey in smokers.The test product should be used for 7 weeks. Seven group meetings are planned during the first 3 months followed bu follow-up sessions after 6 and 12 months. The design is open, randomized. Assessment of ECG, blood pressure, body-weight, carbon monoxide,lung function, stress, quality of life,withdrawal symptoms,adverse events and plasma nicotine, cotinine and thiocyante at entry and after 4 weeks etc.

ELIGIBILITY:
Inclusion Criteria:

* smoking > 13 cigarettes/day
* healthy (allowed: hypertension, diabetes type 2, mild asthma/COPD, hypercholesterolemia)
* motivated for cessation
* motivated to use tobacco pastils
* motivated for group support

Exclusion Criteria:

* severe diseases
* psychiatric diseases
* using antipsychotic drugs
* used NRT/bupropion in the last 3 months
* consuming > 6 drinks/day
* pregnant/lactating
* stopped smoking more than 2 days during last 3 months

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-03; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Continuous Smoking cessation quit rate after 6 and 12 months

SECONDARY OUTCOMES:
Side effects from tested tobacco product
Intake of nicotine and thiocyanate

CONTACTS AND LOCATIONS:
Overall Officials: Philip Tønnesen, M.D., Ph.D., Study Chair — Chair dept. pulm. medicine, Gentofte Hospital
Locations (1):
- Dept. pulmonary medicine Y, Gentofte University Hospital, Copenhagen, Hellerup, Denmark

REFERENCES:
- [Result] Tonnesen P, Mikkelsen K, Bremann L. Smoking cessation with smokeless tobacco and group therapy: an open, randomized, controlled trial. Nicotine Tob Res. 2008 Aug;10(8):1365-72. doi: 10.1080/14622200802238969. PMID 18686184